CLINICAL TRIAL: NCT01962493
Title: A Study to Evaluate the Effect of a 67% Sodium Bicarbonate Containing Toothpaste on Chlorhexidine Digluconate Tooth Staining
Brief Title: An Efficacy Study of Stain Control of a 67% Sodium Bicarbonate Containing Toothpaste on Chlorhexidine Tooth Staining
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202182; RH01913 (Other: GSK)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Fluoride; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sodium bicarbonate/ Sodium Fluoride toothpaste (Other): Marketed Sodium bicarbonate toothpaste containing 1400 parts per million (ppm) fluoride as Sodium fluoride (NaF)
  Interventions: Other: Sodium bicarbonate/ Sodium Fluoride
- Sodium fluoride toothpaste (Active Comparator): Non-sodium bicarbonate toothpaste containing 1450ppm fluoride as NaF
  Interventions: Other: Sodium fluoride
- Chlorhexidine digluconate mouthwash (Other): 0.2% w/v Chlorhexidine digluconate mouthwash for rinsing post-brushing with study toothpastes
  Interventions: Drug: Chlorhexidine digluconate

INTERVENTIONS:
Other: Sodium bicarbonate/ Sodium Fluoride — Toothpaste containing sodium bicarbonate and sodium fluoride as cosmetic
  Arms: Sodium bicarbonate/ Sodium Fluoride toothpaste
Other: Sodium fluoride — Toothpaste containing sodium fluoride as cosmetic
  Arms: Sodium fluoride toothpaste
Drug: Chlorhexidine digluconate — Mouthwash containing chlorhexidine digluconate
  Arms: Chlorhexidine digluconate mouthwash

SUMMARY:
The aim of this study is to compare the stain effect on teeth of twice daily brushing with a 67% sodium bicarbonate containing toothpaste versus standard toothpaste (not containing sodium bicarbonate) for six weeks whilst using a chlorhexidine digluconate 0.2% mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* Good oral health in the opinion of the investigator (excluding gingivitis)
* A minimum of 11 of the 12 permanent gradable anterior teeth at screening
* Stain levels on the buccal surfaces of the 6 maxillary and 6 mandibular anterior teeth need to be at least "mild" and present on a minimum of 4 teeth
* Modification of the Lobene Stain Index - At Visit 2, a baseline total MLSI Intensity x Area score (four sites per tooth) of greater than or equal to 8 for facial surfaces of anterior teeth.

Exclusion Criteria:

* Pregnant women or women who are intending to become pregnant over the duration of the study
* Known or suspected intolerance or hypersensitivity to Chlorhexidine or other study materials (or closely related compounds).
* Current use of Chlorhexidine, Cetylpyridinium Chloride or any marketed mouthwash
* Past or current use of any drug which is known to be associated with tooth discolouration within 30 days of screening or during the study period.
* Recent history (within the last 1 year) of alcohol or other substance abuse
* Dental conditions / disease requiring immediate treatment; Crowns or veneers on more than one anterior tooth; pre-existing sensitivity to oral care products; severe periodontitis; severe recession; dental implants; active carious lesions on anterior teeth; oral lesions/manifestations; prone to aphthous stomatitis and ulceration etc.
* Participant with untreated oral mucosal disease which in the opinion of the investigator could interfere with the study.
* Medical condition which would require the use of prophylactic antibiotics prior to dental cleanings
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder that would make the participant unlikely to fully complete the study or any condition that presents undue risk from the study treatment or procedures in the opinion of the investigator or dental assessor.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - Intertek 4-Front Research - Widnes, Widnes, Cheshire
  - Intertek - Maldon (formerly 4 Front Research Ltd), Maldon, Essex
  - Intertek - Manchester Science Park, Manchester

REFERENCES:
- [Derived] Akwagyiram I, Butler A, Maclure R, Colgan P, Yan N, Bosma ML. A randomised clinical trial to evaluate the effect of a 67 % sodium bicarbonate-containing dentifrice on 0.2 % chlorhexidine digluconate mouthwash tooth staining. BMC Oral Health. 2016 Aug 25;16(1):79. doi: 10.1186/s12903-016-0271-3. PMID 27557865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two sites in the UK. Participants were recruited from the site's database and by use of advertisements.
Pre-assignment Details: In total 314 participants were screened and 160 participants were randomised of whom 150 completed the study. Of the 10 participants that did not completed the study, 3 had adverse events; 1 had protocol violation and 6 had withdrawal of consent.
Groups:
- NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash: Participants applied a strip of 67% Sodium bicarbonate (NaHCO3) toothpaste (containing 1400 parts per million (ppm) fluoride as Sodium fluoride (NaF)) and brushed for one timed minute. After brushing their teeth, participants rinsed their mouths thoroughly with water and waited 5 timed minutes before rinsing with 10 millilitres (mL) of 0.2% w/v Chlorhexidine Digluconate mouthwash for one timed minute in their normal manner.
- NaF Toothpaste + Chlorhexidine Digluconate Mouthwash: Participants applied a strip of Non-sodium bicarbonate toothpaste containing 1450 ppm fluoride as NaF and brushed for one timed minute. After brushing their teeth, participants rinsed their mouths thoroughly with water and waited 5 timed minutes before rinsing with 10 millilitres (mL) of 0.2% w/v Chlorhexidine Digluconate mouthwash for one timed minute in their normal manner.
Period: Overall Study
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Started | 78 | 82
Completed | 73 | 77
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (11.08) | 39.5 (10.87) | 39.6 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 116
  Male | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Modified Lobene Stain Index (MLSI) at Week 6
Description: An assessment of the area and intensity of dental stain on the study teeth was performed using the MLSI after usage of 0.2% w/v chlorhexidine digluconate mouthwash for 6 weeks. The intensity of stain was scored on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Intensity X Area was thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Week 6 post treatment administration
Population: The efficacy analysis was performed on the Intent-to-treat (ITT) population which consisted of all participants who were randomized and received the study treatment and completed one of the post-baseline efficacy assessments.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.97 (0.929) | 1.22 (1.008)
Statistical Analysis 1: Comparison: NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash vs NaF Toothpaste + Chlorhexidine Digluconate Mouthwash; Null hypothesis stated that there was no difference between treatment groups; Test type: Superiority or Other; p = 0.1313, ANCOVA — Analysis based on square root transformation. Results back transformed for interpretation; Results were obtained from ANCOVA model with Site, Treatment, Treatment X Site, Smoking Status as fixed effects and baseline MLSI as a covariate; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.51 to 0.10], Standard Error of Mean 0.155 — Difference is first named treatment minus second named treatment. A negative difference favors the first named treatment

2. Secondary Outcome: Overall MLSI at Week 3
Description: An assessment of the area and intensity of dental stain on the study teeth was performed using the MLSI after usage of 0.2% w/v chlorhexidine digluconate mouthwash for 3 weeks. The intensity of stain was scored on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Intensity X Area was thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Week 3 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.46 (0.572) | 0.59 (0.563)

3. Secondary Outcome: Overall Facial MLSI at Week 3
Description: as for outcome 2
Time Frame: Week 3 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.27 (0.557) | 0.41 (0.542)

4. Secondary Outcome: Overall Facial MLSI at Week 6
Description: as for outcome 1
Time Frame: Week 6 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.67 (0.885) | 0.96 (0.992)

5. Secondary Outcome: Overall Interproximal MLSI at Week 3
Description: as for outcome 2
Time Frame: Week 3 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.66 (0.828) | 0.87 (0.820)

6. Secondary Outcome: Overall Interproximal MLSI at Week 6
Description: as for outcome 1
Time Frame: Week 6 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 1.44 (1.396) | 1.87 (1.525)

7. Secondary Outcome: Overall Gingival and Interproximal MLSI at Week 3
Description: as for outcome 2
Time Frame: Week 3 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 0.56 (0.713) | 0.73 (0.711)

8. Secondary Outcome: Overall Gingival and Interproximal MLSI at Week 6
Description: as for outcome 1
Time Frame: Week 6 post treatment administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Number analyzed (Participants) | 75 | 79
Score on a Scale | 1.18 (1.134) | 1.52 (1.271)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the washout period, and until five days following last administration of the investigational product
Arm/Group | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/82
Other Adverse Events (participants affected / at risk) | 39/78 | 41/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash (N=78) | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash (N=82)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Ruptured Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaHCO3/NaF Toothpaste + Chlorhexidine Digluconate Mouthwash (N=78) | NaF Toothpaste + Chlorhexidine Digluconate Mouthwash (N=82)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 4 (4)
Glossodynia (Gastrointestinal disorders) | 2 (2) | 3 (4)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (3)
Sensitivity of teeth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tongue discolouration (Gastrointestinal disorders) | 4 (4) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 13 (14) | 6 (9)
Dysgeusia (Nervous system disorders) | 1 (1) | 7 (7)
Tension headache (Nervous system disorders) | 4 (6) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 8 (8)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device failure (General disorders) | 1 (1) | 1 (1)
Cyst rupture (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.